CLINICAL TRIAL: NCT04484233
Title: Evaluation of a Clinical Decision Support System for Anemia Management in Pre-operative Care: Feasibility & Validation Study
Brief Title: Evaluation of a Clinical Decision Support System for Anemia Management in Pre-operative Care
Acronym: iAnemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Intelligence Anesthesia (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB 00010254-2020-131
Record Dates: First submitted 2020-07-18; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Decision Support Systems; Anemia
Keywords: Clinical Decision Support Systems; Patient Blood Management; Preoperative Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control Group: Anesthesiologists would have to respond to an online questionnaire about 10 hypotheticals clinical situations regarding patient blood management.
- Clinical Decision Support Group: Anesthesiologists would have to respond to an online questionnaire about 10 hypotheticals clinical situations regarding patient blood management helped by dedicated clinical decision support systems for patient blood management (iAnemia, Intelligence Anesthesia).
  Interventions: Device: iAnemia Decision Support System

INTERVENTIONS:
Device: iAnemia Decision Support System — iAnemia permits to display the appropriate guideline using several inputs about a patient: age, type and delay of the surgery, gender, hemoglobin level, and iron deficiency status.
  Groups: Clinical Decision Support Group

SUMMARY:
Anemia need to be diagnosed and treated, following several guidelines. However, the complexity of these recommendations leads to low compliance and to unnecessary and harmful per- and postoperative blood transfusion.

In order to improve practices and regarding the complexity of the guidelines, the latest European Consensus Conference recommends the use of decision support systems for the management of preoperative anemia.

DETAILED DESCRIPTION:
The World Health Organization defines anemia as a hemoglobin level of less than 13 g/dL in adult men and less than 12 g/dL in women.

The cause of these anemias is most often deficient with 17% iron deficiency. This deficiency is related to age, inflammatory diseases, blood loss, and absorption disorders mainly. Anemia must be diagnosed preoperatively and treated.

To reduce transfusion in the perioperative period there are various possibilities: increase of the preoperative erythrocyte mass, reduction of losses, use of the blood that has been applied.

The impact of these preoperative strategies can be considerable. In their work, Beattie and al demonstrates that transfusion is associated with an increase in mortality at 90 days, proportional to the volume transfused, with certainly a higher risk in fragile subjects. More recently, an American registry of more than 220,000 patients showed that 30% had preoperative anemia. This anemia not only significantly increased mortality, but all causes of comorbidity were aggravated in an anemic patient.

However, the complexity of these recommendations leads to low compliance and to unnecessary and harmful per- and postoperative blood transfusion.

In order to improve practices and regarding the complexity of the guidelines, the latest European Consensus Conference recommends the use of decision support systems for the management of preoperative anemia.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologist: anesthesiologists, resident/fellow physician anesthesiologists.

Exclusion Criteria:

* Unfinished questionnaire.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anesthesiologist:
  * Less than one year experience in anesthesia
  * 2 to 5 years of experience
  * 5 to 10 years of experience
  * 10 to 20 years of experience
  * More than 20 years of experience
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Average global score obtained for the two groups. | Up to 24 weeks
  The mean number of correct answers (out of possible 10);

SECONDARY OUTCOMES:
Average subcategories score obtained for the two groups. | Up to 24 weeks
  The mean number of correct answers (out of possible 10);

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mueller MM, Van Remoortel H, Meybohm P, Aranko K, Aubron C, Burger R, Carson JL, Cichutek K, De Buck E, Devine D, Fergusson D, Follea G, French C, Frey KP, Gammon R, Levy JH, Murphy MF, Ozier Y, Pavenski K, So-Osman C, Tiberghien P, Volmink J, Waters JH, Wood EM, Seifried E; ICC PBM Frankfurt 2018 Group. Patient Blood Management: Recommendations From the 2018 Frankfurt Consensus Conference. JAMA. 2019 Mar 12;321(10):983-997. doi: 10.1001/jama.2019.0554. PMID 30860564
- [Background] Rothschild JM, McGurk S, Honour M, Lu L, McClendon AA, Srivastava P, Churchill WH, Kaufman RM, Avorn J, Cook EF, Bates DW. Assessment of education and computerized decision support interventions for improving transfusion practice. Transfusion. 2007 Feb;47(2):228-39. doi: 10.1111/j.1537-2995.2007.01093.x. PMID 17302768
- [Background] Adams ES, Longhurst CA, Pageler N, Widen E, Franzon D, Cornfield DN. Computerized physician order entry with decision support decreases blood transfusions in children. Pediatrics. 2011 May;127(5):e1112-9. doi: 10.1542/peds.2010-3252. Epub 2011 Apr 18. PMID 21502229